CLINICAL TRIAL: NCT00094341
Title: An Open-Label, Randomized, Crossover Study to Assess Preference of Rheumatoid Arthritis (RA) Patients of Enbrel® (Etanercept) Auto-Injector Versus Enbrel® Pre-Filled Syringes
Brief Title: Preference of Rheumatoid Arthritis (RA) Patients of Enbrel® (Etanercept) Auto-Injector Versus Enbrel® Pre-Filled Syringes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20040201
Record Dates: First submitted 2004-10-16; First posted 2004-10-18 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Arthritis; Rheumatology
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The purpose of this study is to determine the preference of RA patients for the new Enbrel® (etanercept) pre-filled syringe in patients who are already taking Enbrel®.

ELIGIBILITY:
Inclusion Criteria:

* Have established RA diagnosis as determined by ACR criteria
* Be current user of etanercept-lyophilized preparation for at least 4 consecutive weeks of etanercept dosing on either a once weekly or twice weekly regimen
* Subject must be able to self inject
* Give written informed consent

Exclusion Criteria:

* Subject is currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug trial(s), or subject is receiving other investigational agent(s)
* Subject of childbearing potential is pregnant (e.g., positive HCG test) or is breast-feeding
* Elective surgery is planned during study period
* Subjects allergic to latex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215
Dates: Start 2004-10

PRIMARY OUTCOMES:
The proportion of patients preferring the etanercept auto-injector to the etanercept pre-filled syringe.

SECONDARY OUTCOMES:
The proportion of patients preferring the etanercept auto-injector to the etanercept pre-filled syringe as well as to the lyophilized preparation in the following categories:
Ease of use
Hand discomfort during the injection
Satisfaction with number of steps
Time involved with the injection
Nervousness with injection
Confidence with the injection
Convenience of use and
Overall preference with the auto-injector or pre-filled syringes compared to the lyophilized preparation.
To characterize the ability of patients to properly use by themselves either device independently and identify any sections of the instructions that were not clear, that may have led to loss of sterility to incomplete dosing

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: FDA-approved Drug Labeling — http://www.enbrel.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_916_ENBREL_20040201.pdf